CLINICAL TRIAL: NCT00201708
Title: Phase II Randomized Adjuvant Trial of Dose-Dense Docetaxel Before or After Doxorubicin/Cyclophosphamide (AC) in Axillary Node-Positive Breast Cancer
Brief Title: Dose-Dense Docetaxel Before or After Doxorubicin/Cyclophosphamide in Axillary Node-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0450
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Adjuvant Trial; Dose-Dense; Axillary Node-Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Docetaxel before doxorubicin/cyclophosphamide) (Active Comparator): Docetaxel 75 mg/m2 every 2 weeks for 4 cycles followed by "A" (doxorubicin) 60 mg/m2 & "C" (cyclophosphamide) 600 mg/m2 every 2 weeks for 4 cycles.
  Interventions: Drug: Docetaxel; Drug: Doxorubicin; Drug: Cyclophosphamide (AC)
- Arm B (Docetaxel after doxorubicin/cyclophosphamide) (Active Comparator): "A" (doxorubicin) 60 mg/m2 & "C" (cyclophosphamide) 600 mg/m2 every 2 weeks for 4 cycles followed by Docetaxel 75 mg/m2 every 2 weeks for 4 cycles.
  Interventions: Drug: Docetaxel; Drug: Doxorubicin; Drug: Cyclophosphamide (AC)

INTERVENTIONS:
Drug: Docetaxel — Arm A:75 mg/m2 every 2 weeks)for 4 cycles. Arm B:75 mg/m2 every 2 weeks for 4 cycles.
  Other Names: Taxotere
Drug: Doxorubicin — 60 mg/m2 intravenously as push over 2-5 minutes, every 14 days for 4 cycles. Arms: Arm A (Docetaxel before doxorubicin/cyclophosphamide) , Arm B (Docetaxel after doxorubicin/cyclophosphamide)
  Other Names: Adriamycin; hydroxydaunorubicin
Drug: Cyclophosphamide (AC) — 600 mg/m2 over 30 to 60 minutes every 14 days (2 weeks) for 4 cycles. Arms: Arm A (Docetaxel before doxorubicin/cyclophosphamide), Arm B (Docetaxel after doxorubicin/cyclophosphamide)
  Other Names: Cytoxan; CPM; CTX; CYT

SUMMARY:
This study will determine if docetaxel will be administered before or after doxorubicin/cyclophosphamides in an adjuvant chemotherapy regimen to be evaluated in a subsequent phase III trial.

DETAILED DESCRIPTION:
Rationale: Studies suggest that chemotherapy agents docetaxel, doxorubicin, and cyclophosphamide have some efficacy against different types of breast cancer. However, the optimal sequence in which to administer these treatments remains unknown. The current study assesses two separate sequences of docetaxel, doxorubicin, and cyclophosphamide.

Purpose: This study will evaluate two different combination chemotherapy schedules for patients with axillary node-positive breast cancer. Combination one is docetaxel before doxorubicin and cyclophosphamide. Combination two is docetaxel after doxorubicin and cyclophosphamide. The combination with no dose reductions of docetaxel within 10 weeks will then be tested in a Phase III study. The toxicities of docetaxel will also be assessed in study participants.

Treatment: Patients in this study will receive one of two chemotherapy combination schedules. A computer will randomly assign patients into their treatment group. Group one will receive docetaxel before doxorubicin and cyclophosphamide. Group two will receive docetaxel after doxorubicin and cyclophosphamide.

Patients in group one will receive docetaxel every two weeks for a total of eight weeks. These patients will then be given combination doxorubicin and cyclophosphamide every two weeks for a total of eight weeks. Patients in group two will receive combination doxorubicin and cyclophosphamide every two weeks for a total of eight weeks. These patients will then be given docetaxel every two weeks for a total of eight weeks.

Several tests and exams will be given throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed breast cancer
* No metastatic disease
* Prior lumpectomy or mastectomy
* No prior chemotherapy or hormone treatments for breast cancer
* Must have normal organ and marrow function.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.

Exclusion Criteria:

* Peripheral neuropathy of grade II or higher.
* History or evidence upon physical exam of CNS (central nervous system Diseases)disease.
* History of unstable angina or myocardial infarction within the last six months.
* Pregnant or nursing women.
* Known allergies to polysorbate 80.
* HIV-positive patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Select one of two adjuvant chemotherapy regimens for evaluation in subsequent phase III trial. | up to 8 weeks
  Docetaxel before doxorubicin/cyclophosphamide(AC)or Docetaxel after AC. The regimen selection will be based on the proportion of patients receiving four cycles of Docetaxel with no dose reductions within 10 weeks.

SECONDARY OUTCOMES:
Determine the toxicities of Docetaxel administered before or after doxorubicin/cyclophosphamide(AC). | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Shapiro, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Puhalla S, Mrozek E, Young D, Ottman S, McVey A, Kendra K, Merriman NJ, Knapp M, Patel T, Thompson ME, Maher JF, Moore TD, Shapiro CL. Randomized phase II adjuvant trial of dose-dense docetaxel before or after doxorubicin plus cyclophosphamide in axillary node-positive breast cancer. J Clin Oncol. 2008 Apr 1;26(10):1691-7. doi: 10.1200/JCO.2007.14.3941. Epub 2008 Mar 3. PMID 18316792
- See also: Jamesline — http://cancer.osu.edu